CLINICAL TRIAL: NCT06590389
Title: The Effect Of Mandala Activity On Postoperative Pain And Anxiety Levels In Gynecological Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayça Demir Yıldırım, PhD, Assistant Professor, PhD, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAkyol-001
Record Dates: First submitted 2024-07-07; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cancer Pain; Cancer, Treatment-Related; Cancer
Keywords: pain; anxiety; midwife; Gynecological Oncology; mandala
MeSH Terms: conditions — Cancer Pain; Neoplasms, Second Primary; Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research was designed as a randomized controlled, 2-group (intervention and control) pre-test post-test comparative experimental research.
Who Masked: Participant
Masking Description: Randomizer.org website was used for randomization of the research sample. It consists of four rooms, patient room numbers 634, 635, 636 and 637. The room numbers obtained during randomization were assigned to the 1st group intervention (21 cases of open abdominal surgery) and the 2nd group to the control group (21 cases of open abdominal surgery) by simple random method. By entering the room numbers into two unique sets, patients sleeping in the rooms in the 1st set (634-636) and meeting the inclusion criteria were included in the intervention group. Patients sleeping in the rooms in the 2nd set (635-637) and meeting the inclusion criteria were included in the control group. was included in the group. In the study, each patient was included in the research group after informed consent was obtained. In case of refusal, consent was obtained from the next patient in the room and the process of obtaining consent was continued until the number of samples was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Mandala activity) (Experimental): Mandala activity is painting with different pictures or shapes by creating a harmony of figures in different or the same colors. The entire intervention group was given a booklet consisting of 10 simple mandala drawings prepared by the researchers. Mandala activity: During the hospital stay on the zeroth, first and second postoperative days, the patient was asked to color the mandala drawing of his choice from the booklet as many times as he wanted. However, they were asked to practice at least one mandala activity every day. For painting in the mandala activity, a set of 12 colored crayons was given to the patients by the researcher and no color guidance was given for painting. The research was continued by following up within 3 days, namely the zeroth, first and second postoperative days. VAS and STAI-I forms were applied before and after the mandala activity.
  Interventions: Other: mandala activity
- Control group (No Intervention): After the patient was mobilized on the zero postoperative day, STAI-I and VAS were applied 1 hour apart. VAS was repeated every 4 hours until the patient was discharged.
  * On the first day after surgery, VAS with STAI-I was applied to the patient every 1 hour after breakfast, and VAS was repeated every 4 hours during the day.
  * On the second day after the surgery, STAI-I and VAS were applied to the patient 1 hour apart after breakfast.
  * On the second postoperative day, the Postoperative Period Patient Evaluation form was applied to the patient before discharge.

INTERVENTIONS:
Other: mandala activity — A descriptive patient form, VAS and STAI-I were applied before surgery. After the surgery, VAS and STAI-I were applied before and after the mandala activity until the patient was discharged. The VAS form was applied every 4 hours until the patient was discharged. This process was repeated in the same way for the entire intervention group.
  Arms: Intervention group (Mandala activity)

SUMMARY:
This study was designed as a randomised controlled, 2-group, pre-test post-test comparative, experimental study to examine the effect of mandala activity on postoperative pain, anxiety levels and analgesia use of gynaecological oncology patients.

DETAILED DESCRIPTION:
This study was designed as a randomised controlled, 2-group, pre-test post-test comparative, experimental study to examine the effect of mandala activity on postoperative pain, anxiety levels and analgesia use of gynaecological oncology patients.

The study was conducted with 42 patients who underwent open abdominal hysterectomy surgery in the Gynecological Oncology Surgery Clinic of a training and research hospital in Istanbul between 1 February 2023 and 1 August 2023. Patients in the intervention group (n=21) received mandala activity at least once a day during their postoperative hospitalisation (days 0-2). Patients in the control group (n=21) did not receive any intervention. Introductory Information Form, Visual Analogue Scale (VAS), State-Trait Anxiety Inventory (STAI-I), Postoperative Patient Evaluation Form and Mandala Activity Booklet were used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Having a gynecological oncology disease diagnosis,
* Having had open abdominal hysterectomy surgery,
* Being over 18 years of age,
* Ability to communicate in Turkish,
* Having a gynecological oncology operation for the first time,
* There is no physical disability related to the upper extremities.

Exclusion Criteria:

* Readmission due to any complications that develop after discharge,
* Having visual, hearing and speech disabilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with gynecological oncology disease
Enrollment: 42 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1 February 2023 - 1 August 2023 (6 months or 182 days)
  This scale is used to visually assess and then quantify values that cannot be measured quantitatively. It was used to measure the pain intensity of gynecologic oncology patients in both the intervention and control groups. In this scale, the variable to be evaluated is written on both ends of a 100 mm long line. The patient was asked to place a line, dot or cross on this beam by asking which one she was closer to. For example, the leftmost part is labeled "no pain" and the other end is labeled "most severe pain". The patient makes a mark on the ray according to his/her current condition. Starting from the left end, i.e. where there is no pain at all, the part up to the point where the patient has pain, i.e. where the patient makes a mark, is measured. This quantity indicates the intensity of the patient's pain. The increase in quality and quantity indicates an increase in pain intensity.

SECONDARY OUTCOMES:
Number of analgesia use | 1 February 2023 - 1 August 2023 (6 months or 182 days)
  It is a form used to evaluate the use of postoperative analgesia in gynaecological oncology patients.

OTHER OUTCOMES:
State-Trait Anxiety Inventory I (STAI-I) | 1 February 2023 - 1 August 2023 (6 months or 182 days)
  The scale measures state and trait anxiety as Likert scale with 20 separate questions. The higher the scores, the higher the level of anxiety and the lower the scores, the lower the level of anxiety. The total score of both scales ranges from a minimum of 20 to a maximum of 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Demir Yıldırım, Phd, Study Director — https://uskudar.edu.tr/akademik-personel/ayca-demir-yildirim
Locations (1):
- Üsküdar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A research paper was planned to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] T.C. Ministry of Health Public Health Institution of Turkey 2013-2018 National Cancer Control Plan, Ed: Keskinkılıç B. [Internet]. 2022 [Accessed on 3.10.2022]. Access address: https://hsgm.saglik.gov.tr/depo/birimler/kanser-db/yayinlar/raporlar
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] TÜİK. Cause of Death Statistics, 2017. tuikweb.tuik.gov.tr/PreHaberBultenleri.do?id=27592 https://hsgm.saglik.gov.tr/depo/birimler/kanser-db/istatistik/Turkiye_Kanser_Istatistikleri_2017.pdf Date of access: 1.10.2022
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Hawkins Y, Ussher J, Gilbert E, Perz J, Sandoval M, Sundquist K. Changes in sexuality and intimacy after the diagnosis and treatment of cancer: the experience of partners in a sexual relationship with a person with cancer. Cancer Nurs. 2009 Jul-Aug;32(4):271-80. doi: 10.1097/NCC.0b013e31819b5a93. PMID 19444088
- [Background] Afiyanti Y, Milanti A, Putri RH. Supportive care needs in predicting the quality of life among gynecological cancer patients. Can Oncol Nurs J. 2018 Feb 1;28(1):22-29. doi: 10.5737/236880762812229. eCollection 2018 Winter. PMID 31148629
- [Background] Jiang XH, Chen XJ, Xie QQ, Feng YS, Chen S, Peng JS. Effects of art therapy in cancer care: A systematic review and meta-analysis. Eur J Cancer Care (Engl). 2020 Sep;29(5):e13277. doi: 10.1111/ecc.13277. Epub 2020 Jun 15. PMID 32542749
- [Background] Spielberger, C. D. (1983). State-trait anxiety inventory for adults. Mind Garden.https://www.tandfonline.com/doi/pdf/10.1080/07481756.1985.12022795